CLINICAL TRIAL: NCT04522882
Title: Development of a Closed Loop for the Treatment of Type 2 Diabetes: Collection of Clinical Data at Home for the Creation of an Algorithmic Laboratory Test Bench
Brief Title: Clinical Data Collection for the Closed Loop Development for the Type 2 Diabetes Treatment - DT2_1
Acronym: DT2_1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diabeloop (Industry)
Collaborators: Icadom (Industry); AGIR à Dom (Other); CHU Grenoble Alpes (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RCB 2020-A01710-39
Record Dates: First submitted 2020-07-23; First posted 2020-08-21 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2020-09

CONDITIONS: Type 2 Diabetes Treated With Insulin
Keywords: Type 2 diabetes; Insulin; Life conditions; Algorithm; Closed loop
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Actimetry is performed in all patients included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- At home clinical data collection (Experimental): Clinical data will be collected during 7 days: physical activity, sleep duration, chronotype, food and medication intake, glucose level and insulin administration.
  Interventions: Device: Actimetry; Other: Questionnaires; Other: Glucose level and insulin administration

INTERVENTIONS:
Device: Actimetry — Actimetry will be performed at home to measure physical activity, sleep duration and patient chronotype for 7 days.
Other: Questionnaires — Patients will complete food and medication intake questionnaires for 7 days.
Other: Glucose level and insulin administration — Continuous subcutaneous glucose level (measured by continuous glucose monitor (CGM)) and the insulin doses delivered by the insulin pump will be collected for 7 days .

SUMMARY:
The objective of this study is to collect the evolution of blood glucose levels in type 2 diabetes (T2D) patients under different conditions of their daily life: physical activity, meals, sleep, etc. This data will be used to develop a test bench to evaluate insulin delivery algorithms to treat patients with insulin-resistant T2D using a closed loop.

DETAILED DESCRIPTION:
T2D is a condition that combines insulin resistance and relative insulin deficiency. The T2D naturally progresses towards an increasingly pronounced insulin deficiency that leads to the need for pancreatic replacement, by administering insulin.

Type 1 diabetes (T1D) requires a complete and immediate substitution of pancreatic insulin secretion. Currently, patients need to be involved in managing their disease by deciding how much insulin to administer based on the results of glucose monitoring. Artificial intelligence, thanks to a self-learning algorithm, enables the automation and customization of insulin administration. These devices, known as closed loops, bring real benefit to the patients included in the studies, by improving glycemic balance, by decreasing the number of hypo- and hyperglycemia but also by decreasing the mental load associated with the disease, improving their quality of life.

These very significant benefits in the T1D treatment open the possibility of obtaining similar benefits in the T2D treated by the basal-bolus type insulin regimen. This study aims to develop a specific algorithm of T2D to meet its particular characteristics.

The objective of this study is to collect the evolution of blood glucose levels in T2D patients under different conditions of their daily life: physical activity, meals, sleep, etc. This data will be used to develop a test bench to evaluate insulin delivery algorithms to treat patients with insulin-resistant T2D using a closed loop.

ELIGIBILITY:
Inclusion Criteria:

* Patient with T2D treated with insulin pump for at least 6 months
* Patient with a body mass index (BMI) between 27 and 40 kg/m2
* Patient treated with a total daily dose of insulin between 40 and 300 U/24 h
* Patient with CGM
* Patient with Social security or beneficiary
* Patient able to read and understand the procedure, and able to express consent for the study protocol

Exclusion Criteria:

* Patient with T1D
* Patient currently participating or having participated in the month prior to inclusion in another interventional clinical research that may impact the study, this impact is left to the investigator's discretion
* Persons referred to in articles L.1121-5 to L.1121-8 of the CSP (corresponds to all the protected persons: pregnant woman (checked by the dosage of β-human chorionic gonadotropin for any woman wishing to participate in the protocol and in childbearing age 60 years), parturient, mother breastfeeding, person deprived of liberty by judicial or administrative decision, person subject to a legal protection measure)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Glucose level modification | 7 days
  Continuous subcutaneous glucose level (measured by continuous glucose sensor (CGM)) for 7 days, compared to the daily activities collected and the insulin doses delivered by the insulin pump.

SECONDARY OUTCOMES:
Physical activity | 7 days
  Measured by actimetry
Physical activity | 7 days
  Measured by physical actimetry journal
Sleep duration | 7 days
  Measured by actimetry
Sleep duration | 7 days
  Measured by sleep journal
Patient's chronotype | 7 days
  Measured by actimetry
Patient's chronotype | 7 days
  Measured by sleep journal
Schedule and type of food intake | 7 days
  Questionnaire on schedule and type of food intake (without score on a scale)
Medication intake | 7 days
  Questionnaire on medication intake (without score on a scale)

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Laure BOREL, MD, PhD, Principal Investigator — CHU Grenoble Alpes
Locations (1):
- AGIRADOM, Meylan, France

IPD SHARING:
Plan to Share IPD: No